CLINICAL TRIAL: NCT05118373
Title: Evaluation of a Generic Behavioural Change Campaign for COVID-19 Prevention in Zambia
Brief Title: Generic Behavioural Change Campaign for COVID-19 Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25741
Record Dates: First submitted 2021-08-18; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Evaluation Study
Keywords: Behavioural change, Evaluation, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Nation-wide mass media behaviour change campaign.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure (Other): The campaign targets 3 TV stations, 8 radio stations, 2 billboard companies and social media platforms including YouTube, Twitter, Facebook, Instagram and LinkedIn with an anticipated reach of 1,433,201 people in Lusaka and Copperbelt provinces. Of the targeted TV and radio media houses, two each are national stations and will reach beyond these two intervention provinces including to Central and Southern province with an estimated 8% and 11% mass-media penetration compared to 21% and 38% for Copperbelt and Lusaka respectively.
  Interventions: Behavioral: BEHAVIOURAL CHANGE CAMPAIGN FOR COVID-19 PREVENTION IN ZAMBIA

INTERVENTIONS:
Behavioral: BEHAVIOURAL CHANGE CAMPAIGN FOR COVID-19 PREVENTION IN ZAMBIA — The intervention is a mass media campaign using TV, radio, billboard and posters to disseminate the message. The content are well-produced videos and pictures emphasising the need to wash hands, wear a mask, maintain social distance and clean surfaces. The English version of the video can be viewed at this link: https://youtu.be/tcjaLAxy4Ms.

SUMMARY:
Since the start of the COVID-19 pandemic in Zambia, multiple information, education and communication (IEC) materials and strategies have been disseminated by national risk communication and community engagement (RCCE) committees to create awareness on the facts of the novel coronavirus, prevention measures and care-seeking options. To complement these efforts in Zambia, CIDRZ in collaboration with the London School of Hygiene and Tropical Medicine (LSHTM) are implementing an internationally produced communication campaign that promotes the uptake of four key behaviours to reduce the transmission of COVID-19, namely, hand washing with soap, mask wearing, social distancing and surface cleaning. The campaign presents these behaviours as a 'password' that should be enacted to get lives back to normal and was created by the Hygiene Behaviour Change Coalition (HBCC). The idea of a password has been used to symbolize access into a world where protective habits are practiced in order to get back a world that is corona free. The password in this case is Hands-Face-Space-Surface. This campaign is a mass media campaign that will be delivered through TV, radio and billboards.

This study aims to evaluate the process and effect of the HBCC campaign on the uptake of COVID-19 preventative behaviours among people living in Lusaka and Copperbelt Provinces of Zambia.

DETAILED DESCRIPTION:
Currently, there is not enough evidence on the impact of specific behavioural interventions on the uptake of COVID-19 prevention behaviours, including in Zambia.

The password campaign is rooted in behaviour change principles and was carefully created by the HBCC as a unifying intervention promoting memorability and behaviour uptake. It is being implemented in countries in Asia and Africa to increase the uptake of hand washing with soap, mask wearing, social distancing and surface cleaning. This study will be the first to provide evidence on the impact of this intervention on the uptake of behaviours within low-resourced settings.

Research questions:

1. To what extent have adults aged 18years and above been exposed to the password campaign?
2. What effect has the HBCC campaign had on practice of COVID-19 prevention behaviours in the community?

Main Aim: This study aims to evaluate the process and effect of the HBCC campaign on the uptake of COVID-19 preventative behaviours among people living in Lusaka and Copperbelt Provinces of Zambia.

Specific objectives:

1. To assess the contribution of process indicators on the performance of the HBCC campaign with respect to dose delivered and reach.
2. To evaluate the effect of the HBCC campaign on COVID-19 preventative behaviours.

Methodology (design, sampling, data collection methods and tools): In order to assess the intervention effect of the HBCC mass media campaign on the uptake of COVID-19 prevention behaviours among the general population, we will use a post-test quasi-experimental design where we will compare the uptake of three COVID-19 prevention behaviours among the general population in four provinces (Lusaka, Copperbelt, Southern and Eastern), where the intervention is variably ongoing. We will compare responses between exposed to unexposed individuals after intervention (i.e., a per protocol analysis). We define exposure as a positive response about exposure to, and memory of, the Password campaign (in particular it's specific slogan). We will stratify on biological sex and age.

Interactive Voice Response (IVR), an automated telephone system technology that interacts with the callers and routes the calls to the appropriate recipient will be used to collect data. This method had been chosen due to restriction on face to face data collection as a result of the COVID-19 pandemic. A random sample will be drawn from the phone number pool of persons >18 years old registered to participate in surveys.

Data management issues (data management plan, analysis and storage):

Viamo (https://viamo.io/) will provide descriptive analysis for all variables including all respondents. They will further extract fully completed questionnaires and export it to Microsoft excel for cleaning and coding. They will send this de-identified data to CIDRZ, who will export the cleaned data to Stata 16 MP4 (Stata Corp, College Station, TX. USA) for further analyses. De- identification will protect confidentiality. When all the data has been extracted, it will be stored in a database using PostgreSQL object-relational database management for security purposes. PostgreSQL is a highly secure and easy to use.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18years and above
* Must reside in Lusaka, Copperbelt, Southern or Eastern Province
* Volunteer to take part in the study

Exclusion Criteria:

* Participants not from Lusaka, Copperbelt, Southern or Eastern Province

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Behaviour Change | Two months of intervention
  Difference in proportion reporting one of three behaviors (masking, distancing and hand washing among those exposed and not exposed to the mass media campaign

SECONDARY OUTCOMES:
Effective Reach | Two months
  The proportion of people exposed to the intervention who can recall the password
Reach | Two months
  The total number of different people exposed to the intervention, at least once, to any one medium during the two months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anwar A, Malik M, Raees V, Anwar A. Role of Mass Media and Public Health Communications in the COVID-19 Pandemic. Cureus. 2020 Sep 14;12(9):e10453. doi: 10.7759/cureus.10453. PMID 33072461
- [Background] Adewuyi, E. O., 2016. Behavior Change Communication Using Social Media: A Review. THE INTERNATIONAL JOURNAL OF COMMUNICATION AND HEALTH, January.pp. 109-116.
- [Background] Abdullahi L, Onyango JJ, Mukiira C, Wamicwe J, Githiomi R, Kariuki D, Mugambi C, Wanjohi P, Githuka G, Nzioka C, Orwa J, Oronje R, Kariuki J, Mayieka L. Community interventions in Low-And Middle-Income Countries to inform COVID-19 control implementation decisions in Kenya: A rapid systematic review. PLoS One. 2020 Dec 8;15(12):e0242403. doi: 10.1371/journal.pone.0242403. eCollection 2020. PMID 33290402
- [Background] CDC, 2012. Efforts to Prevent and Reduce Tobacco Use Among Young People., Atlanta GA: s.n.
- [Background] Curtis V, Dreibelbis R, Sidibe M, Cardosi J, Sara J, Bonell C, Mwambuli K, Ghosh Moulik S, White S, Aunger R. How to set up government-led national hygiene communication campaigns to combat COVID-19: a strategic blueprint. BMJ Glob Health. 2020 Aug;5(8):e002780. doi: 10.1136/bmjgh-2020-002780. PMID 32764128
- [Background] Graffigna G, Bosio C, Savarese M, Barello M, Barello S. "#I-Am-Engaged": Conceptualization and First Implementation of a Multi-Actor Participatory, Co-designed Social Media Campaign to Raise Italians Citizens' Engagement in Preventing the Spread of COVID-19 Virus. Front Psychol. 2020 Nov 5;11:567101. doi: 10.3389/fpsyg.2020.567101. eCollection 2020. PMID 33250811
- [Background] Lin Y, Hu Z, Alias H, Wong LP. Influence of Mass and Social Media on Psychobehavioral Responses Among Medical Students During the Downward Trend of COVID-19 in Fujian, China: Cross-Sectional Study. J Med Internet Res. 2020 Jul 20;22(7):e19982. doi: 10.2196/19982. PMID 32584779
- [Background] Li X, Liu Q. Social Media Use, eHealth Literacy, Disease Knowledge, and Preventive Behaviors in the COVID-19 Pandemic: Cross-Sectional Study on Chinese Netizens. J Med Internet Res. 2020 Oct 9;22(10):e19684. doi: 10.2196/19684. PMID 33006940
- [Background] Wakefield MA, Loken B, Hornik RC. Use of mass media campaigns to change health behaviour. Lancet. 2010 Oct 9;376(9748):1261-71. doi: 10.1016/S0140-6736(10)60809-4. PMID 20933263
- See also: WASH Matters — http://washmatters.wateraid.org/sites/g/files/jkxoof256/files/wateraids-hygiene-behaviour-change-response-to-covid-19.pdf
- See also: Zambia Risk Communication and Community Engagement — http://reports.unocha.org/en/country/zambia/card/7kSBtUsPLF
- See also: WHO Social Distancing — http://www.who.int/westernpacific/emergencies/covid-19/information/physical-distancing